CLINICAL TRIAL: NCT02973802
Title: Safety and Proof of Principle Study of ATX-GD-59 in Male and Female Subjects With Graves' Disease Not Currently Treated With Anti-thyroid Therapy: An Open Label Study, With an Upward Titration Over Five Dose Levels Administered by Intradermal Injection
Brief Title: ATX-GD-59 in Patients With Graves Disease Not Treated With Anti-thyroid Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Apitope International NV (Industry)
Collaborators: Quintiles, Inc. (Industry); European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATX-GD-59-001
Record Dates: First submitted 2016-11-14; First posted 2016-11-25 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-03

CONDITIONS: Graves Disease
Keywords: Graves Disease; Phase 1
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ATX-GD-59 treatment (Experimental): An upward titration over five dose levels (25, 50, 100, 400 and 800 micrograms) followed by 5 doses of 800 micrograms of ATX-GD-59 will be administered two weeks apart by intradermal injection.
  Interventions: Biological: ATX-GD-59

INTERVENTIONS:
Biological: ATX-GD-59 — Disease specific immune modulating treatment for Graves Disease

SUMMARY:
Phase 1 study to assess the safety and biological activity of ATX-GD-59 in patients with Graves Disease not currently treated with anti-thyroid therapy. This will be an open label dose titration involving injections on 10 occasions, each two weeks apart. After dosing is complete there will be a 12 week follow up period. Blood samples will be drawn throughout the study to monitor safety and the body's response to the injections. Thyroid function will be measured throughout the trial to monitor Graves disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of Graves' disease as assessed by a physician from clinical and laboratory findings and not receiving anti-thyroid therapy.
2. Quantifiable levels of TSHR antibodies.
3. Raised levels of free T3 and/or free T4 (not exceeding 15 pmol/L and 35 pmol/L respectively) including undetectable levels of thyroid stimulating hormone.
4. HLA-DRB1*15, HLA DRB1*03 and or HLA DRB1*04 positive.
5. Age 18 - 65 years inclusive at the time of informed consent.
6. The subject must be willing and able to give written informed consent and must be willing to comply with protocol assessments/procedures.
7. Male subjects must be sterile (biologically or surgically) or commit to the use of a reliable method of birth control for the duration of the study until at least 90 days after the last dose of ATX-GD-59.
8. Female subjects of child bearing potential must: - neither be pregnant nor breast-feeding, nor attempting to conceive, and - use a highly effective method of contraception as defined below, throughout the entire duration of the study and for at least 90 days after the last dose of ATX-GD-59. A serum pregnancy test will be performed at the screening visit in women of child bearing potential. Thereafter urine pregnancy tests will be performed. A positive result will exclude the woman from the study immediately. A highly effective method of contraception is defined as those which result in a low failure rate when used consistently and correctly such as implants, injectable, combined oral contraceptives, some Intrauterine Devices (IUDs), unless post-menopausal or surgically sterilized. Barrier forms of contraception are considered appropriate when used in combination with one of the above methods.

Exclusion Criteria:

1. Subjects who are pregnant or breastfeeding and/or subjects in the post-partum period.
2. A known history of, or hypersensitivity reactions that in the opinion of the investigator would exclude the subjects' participation in the study.
3. Treatment with any Anti-Thyroid Drugs eg carbimazole within the previous 3 months prior to Study Day 1.
4. Previous treatment with radioiodine or (partial or complete) thyroidectomy.
5. Signs of moderate or severe orbitopathy including optic nerve compression requiring steroids and/or a clinical activity score >3.
6. Large and compressive goitres causing localised symptoms such as difficulty swallowing or breathing.
7. Treatment with steroids (administered via the oral and/or parenteral routes) or adrenocorticotropic hormone with the exception of inhaled steroids within the three months prior to Study Day 1.
8. Symptoms and signs of thyroid storm such as confusion, pyrexia with no other cause than hyperthyroidism.
9. Significant cardiac disease and/or atrial fibrillation that would require urgent treatment of thyrotoxicosis.
10. Prior treatment with biological or peptide-based therapeutics including rituximab.
11. Prior use of disease related T cell vaccine or peptide-tolerising agent to treat Graves' disease.
12. Detectable levels of antibodies in plasma specific for any of the peptides within ATX-GD-59 at the screening visit.
13. A history of significant drug allergies.
14. The use of any investigational drug, or participation in any Clinical Trial within three months prior to Study Day 1.
15. Treatment with any cytokine or anti-cytokine therapy within three months prior to Study Day 1.
16. Inadequate liver function, defined by a total bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT) or alkaline phosphatase > 3 times the upper limit of the normal values at Screening visit. 17. Subject with any significant medical illness or psychiatric condition that in the opinion of the Investigator, would preclude participation in the study or impair the ability to give informed consent; any other clinically apparent autoimmune disease.

18. Clinically significant illness, as determined by the investigator, within 4 weeks prior to the first dose (Study Day 1) of ATX-GD-59.

19. Known history of active or chronic infectious disease or any disease which compromises immune function (e.g. HIV+, HTLV-1, Lyme disease, Latent or active TB, Hepatitis).

20. Major surgery in previous four weeks before screening visit. 21. Known osteoporosis or metabolic bone disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon HS Pearce, Principal Investigator — Royal Victoria Infirmary
Locations (8):
- United Kingdom (8):
  - Queen Elizabeth Hospital, Birmingham
  - University Hospital of Wales, Cardiff
  - Royal Devon and Exeter Hospital, Exeter
  - St James's University Hospital, Leeds
  - Hammersmith Hospital, London
  - Kings College Hospital, London
  - The Christie, Manchester
  - Royal Victoria Infirmary, Newcastle

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients diagnosed with Graves Disease from 8 hospital clinics located in the UK. The last patient enrolled completed dosing in February 2018.
Pre-assignment Details: 28 subjects were screened for the study, of which 12 were eligible, and commenced treatment with ATX-GD-59.
Groups:
- ATX-GD-59 Treatment: An upward titration over five dose levels (25, 50, 100, 400 and 800 micrograms) followed by 5 doses of 800 micrograms of ATX-GD-59 administered two weeks apart by intradermal injection.
  ATX-GD-59: Disease specific immune modulating treatment for Graves Disease
Period: Overall Study
Arm/Group | ATX-GD-59 Treatment
Started | 12
Completed | 10
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | ATX-GD-59 Treatment
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11
  Asian | 1

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Treatment Emergent Adverse Events (TEAE), Serious Adverse Events (SAE), and Laboratory Abnormalities up to Week 22 Compared to Baseline.
Description: An adverse event (AE) was defined as any untoward medical occurrence in a subject administered study drug that did not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavourable and unintended sign, symptom, disease or outcome of death temporally associated with the use of study drug, whether or not considered causally related to the study drug. Treatment emergent adverse events (TEAEs) were any AE that started or worsened in severity on or after the first administration of study drug up to and including 28 days after the last administration of study drug. Relationship, as indicated by the Investigator, was classified as 'not related', 'possibly related', 'probably related' or 'definitely related' (increasing severity of relationship). A drug related AE was defined as an AE with a relationship to study drug of 'possibly related', 'probably related' or 'definitely related' or with a missing or unknown relationship to study drug
Time Frame: 22 weeks
Population: The Intention-to-treat population corresponded to all subjects who received at least 1 administration of study drug at any time during the study, irrespective of compliance with eligibility and other protocol criteria. The Safety population was denoted as the 'Intention-to-treat population' for the summarisation of safety endpoints.
Measure: Number; unit: Adverse Events
Arm/Group | ATX-GD-59 Treatment
Number analyzed (Participants) | 12
Adverse Events
  Total Adverse Events | 311
  Mild Adverse Events | 293
  Moderate Adverse Events | 18
  Severe Adverse Events | 0
  Drug Related Adverse Events | 180
  Total Serious Adverse Events | 3
  Drug Related Serious Events | 1
  Adverse Events leading to death | 0
  Adverse Events leading to early study withdrawal | 0
  Events leading to dose interruption or suspension | 0
  Treatment emergent injection related reaction | 153

2. Secondary Outcome: Change in Serum Anti-TSHR Antibodies From Baseline to Week 22 - Measured by TSHR-binding Inhibitory Immunoglobulin (TBII)
Description: TSHR-binding inhibitory immunoglobulin (TBII) are autoantibodies directed against the TSH receptor. TBII is used clinically for the differential diagnosis and management of Graves' Disease.
Time Frame: Weeks 18, 22 and 30
Population: The Intention-to-treat population corresponded to all subjects who received at least 1 administration of study drug at any time during the study, irrespective of compliance with eligibility and other protocol criteria.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | ATX-GD-59 Treatment
Number analyzed (Participants) | 12
IU/L
  Change from baseline at week 18 | -0.7737 (1.55475)
  Change from baseline at week 22 | -0.6602 (1.35220)
  Change from baseline at week 30 | -0.8971 (1.67639)

3. Secondary Outcome: Change in Serum Anti-TSHR Antibodies From Baseline to Week 22 - Measured by Stimulatory TSHR Antibodies (TSAb)
Description: Stimulatory TSHR antibodies (TSAb) assays were measured using cell-based methods described by Leschik et al.
  TSAb activity is measured by calculating percentage specimen-to-reference ratio (%SRR).
Time Frame: Weeks 18, 22 and 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: %SRR
Arm/Group | ATX-GD-59 Treatment
Number analyzed (Participants) | 12
%SRR
  Change from baseline at week 18 | -92.7 (145.73)
  Change from baseline at week 22 | -54.0 (118.94)
  Change from baseline at week 30 | -39.3 (125.36)

4. Secondary Outcome: Change in Serum Anti-TSHR Antibodies From Baseline to Week 22 - Measured by Blocking TSHR Antibodies (TBAb)
Description: Blocking TSHR antibodies (TBAb) assays were measured using cell-based methods described by Leschik et al.
  TBAb activity is measured by calculating percentage inhibition.
Time Frame: Weeks 18, 22 and 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % Inhibition
Arm/Group | ATX-GD-59 Treatment
Number analyzed (Participants) | 12
% Inhibition
  Change from baseline at week 18 | 12.9 (46.50)
  Change from baseline at week 22 | 7.0 (55.54)
  Change from baseline at week 30 | -0.1 (60.49)

5. Secondary Outcome: Change in Serum Free Triiodothyronine (fT3) From Baseline to Week 22.
Description: Serum fT3 was measured centrally from screening to the final week 30 follow-up visit. Baseline was fT3 value at study day 1.
Time Frame: Weeks 18, 22 and 30
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Standard Deviation); unit: Percent change
Arm/Group | ATX-GD-59 Treatment
Number analyzed (Participants) | 12
Percent change
  Change from baseline at week 18 | -11.75 (26.513)
  Change from baseline at week 22 | -14.19 (25.549)
  Change from baseline at week 30 | -15.79 (27.367)

6. Secondary Outcome: Change in Serum Free Thyroxine (T4) From Baseline to Week 22.
Description: Serum fT4 was measured centrally from screening to the final week 30 follow-up visit. Baseline was fT4 value at study day 1.
Time Frame: Weeks 18, 22 and 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | ATX-GD-59 Treatment
Number analyzed (Participants) | 12
Percent change
  Change from baseline at week 18 | -9.80 (24.622)
  Change from baseline at week 22 | -14.54 (20.011)
  Change from baseline at week 30 | -9.24 (27.368)

7. Secondary Outcome: Change in Serum Thyroid Stimulating Hormone (TSH) From Baseline to Week 22.
Description: Serum TSH was measured centrally from screening to the final week 30 follow-up visit. Baseline was fT4 value at study day 1.
Time Frame: Weeks 18, 22 and 30
Population: The Intention-to-treat population corresponded to all subjects who received at least 1 administration of study drug at any time during the study, irrespective of compliance with eligibility and other protocol
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | ATX-GD-59 Treatment
Number analyzed (Participants) | 12
mIU/L
  Change from baseline at week 18 | 0.267 (0.8028)
  Change from baseline at week 22 | 0.309 (0.8398)
  Change from baseline at week 30 | 0.473 (1.1915)

8. Secondary Outcome: Change From Baseline in Peripheral Blood Mononuclear Cell (PBMC) T Cell Activity
Time Frame: weeks 0, 18 and 22
Population: No clear treatment effects could be determined possibly due to technical issues with the preparation and assay of the PBMCs. In addition, the 2 week post dose time point of blood sampling, meant that the induced Treg cells or cytokine changes were no longer detectable in peripheral blood.
Arm/Group | ATX-GD-59 Treatment
Number analyzed (Participants) | 0

9. Secondary Outcome: Change From Baseline in IL-10 mRNA Expression in PBMCs
Time Frame: weeks 0, 18 and 22
Population: as for outcome 8
Arm/Group | ATX-GD-59 Treatment
Number analyzed (Participants) | 0

10. Secondary Outcome: Change From Baseline in Biomarker Signature of PBMC Cells
Time Frame: weeks 0, 18 and 22
Population: as for outcome 8
Arm/Group | ATX-GD-59 Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from screening through to the final follow up visit at week 30.
Description: Adverse events were defined as per clinicaltrials.gov definitions. Adverse events were recorded by investigators and subjects in diaries which were reviewed at each visit. All SAEs and treatment emergent AEs are listed here.
Groups:
- Treatment Emergent Adverse Events: Treatment emergent adverse events were any adverse events that started or worsened in severity on or after the first administration of study drug up to and including 28 days after the last administration of ATX-GD-59
- Non Treatment Emergent Adverse Events: Any non-treatment emergent adverse events.
Arm/Group | Treatment Emergent Adverse Events | Non Treatment Emergent Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 11/12 | 4/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Emergent Adverse Events (N=12) | Non Treatment Emergent Adverse Events (N=12)
Mild Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paroxysmal Atrial Fibrillationion (Cardiac disorders) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Emergent Adverse Events (N=12) | Non Treatment Emergent Adverse Events (N=12)
Injection site erythema (General disorders) | 10 (61) | 0 (0)
Injection site swelling (General disorders) | 8 (46) | 0 (0)
Injection site pain (General disorders) | 6 (27) | 0 (0)
Injection site pruritus (General disorders) | 3 (7) | 0 (0)
Injection site rash (General disorders) | 2 (2) | 0 (0)
Injection site urticaria (General disorders) | 2 (9) | 0 (0)
Pyrexia (General disorders) | 2 (12) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 1 (3) | 0 (0)
Injection site discomfort (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (9) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Suprapubic Pain (General disorders) | 1 (1) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (10) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (13) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 1 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (19) | 0 (0)
Headache (Nervous system disorders) | 3 (10) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibulation (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (4) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0)
Lymph node palpable (Investigations) | 1 (1) | 0 (0)
Respiratory rate increased (Investigations) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Possible Loss of Consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT02973802/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT02973802/SAP_001.pdf